CLINICAL TRIAL: NCT02661776
Title: The Change of NK Cell Activity After Head and Neck Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0987
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: The Patients Undergoing Head and Neck Surgery Including Tumor Removal and Reconstruction With Flap
Keywords: natural killer cell; head and neck cancer; opioid
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood obtained from enrolled patients before and after surgery
Oversight: Data Monitoring Committee: No

SUMMARY:
Cellular immunity can be changed after surgery and anesthesia. Tissue injury by surgical procedures significantly reduces the immune function in proportion to the degree of tissue injury. In addition, the use of opioids as analgesics during the perioperative period depress cellular immunity, in particular the activity of the natural killer (NK) cells. This perioperative immunosuppression may cause deleterious consequences on postoperative outcome in cancer patients. The aim of this study is to confirm the presence or extent of the change of NK cell activity between before and after head and neck surgery. Additionally, investigators will identify the clinical or genetic factors related to the change of NK cell activity.

ELIGIBILITY:
Inclusion Criteria:

1) The patients undergoing head and neck surgery including tumor removal and reconstruction with flap

Exclusion Criteria:

1. patients refusal
2. patients not able to read, or understand the consent form
3. History of Active viral or bacterial infection
4. History of use of immunosuppressive drugs within the last six months
5. History of chemotherapy
6. History of autoimmune disorders
7. Known HIV, Hepatitis B, or Hepatitis C infection
8. Female who is pregnant, nursing
9. ethnicity, other than asian

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing head and neck surgery
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
The change of NK cell activity | 24 hours
  Preoperative NK cell activity will be measured using the NK vue diagnostic test before surgery and anesthesia. Postoperative NK cell activity will be measured using the NK vue diagnostic test after 24 hours since stopping the use of intravenous remifentanil as analgesics during anesthesia in the operating room or sedation in the intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD

REFERENCES:
- [Background] Lee SB, Cha J, Kim IK, Yoon JC, Lee HJ, Park SW, Cho S, Youn DY, Lee H, Lee CH, Lee JM, Lee KY, Kim J. A high-throughput assay of NK cell activity in whole blood and its clinical application. Biochem Biophys Res Commun. 2014 Mar 14;445(3):584-90. doi: 10.1016/j.bbrc.2014.02.040. Epub 2014 Feb 18. PMID 24561245